CLINICAL TRIAL: NCT02510300
Title: A Long Term Follow-up Registry for Adolescent and Pediatric Subjects Who Received a Gilead Hepatitis C Virus Direct Acting Antiviral (DAA) in Gilead-Sponsored Chronic Hepatitis C Infection Trials
Brief Title: A Registry for Adolescent and Pediatric Participants Who Received a Gilead Hepatitis C Virus Direct Acting Antiviral (DAA) in Gilead-Sponsored Chronic Hepatitis C Infection Trials
Status: Terminated | Type: Observational
Why Stopped: The study stopped early because the study objectives were met.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-334-1113; 2014-004674-42 (EudraCT Number)
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir; ledipasvir, sofosbuvir drug combination; velpatasvir; sofosbuvir-velpatasvir drug combination; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sofosbuvir (SOF) — Exposure of interest for participants who received a SOF-based regimen in previous Gilead-sponsored chronic hepatitis C infection trials
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: Ledipasvir/Sofosbuvir (LDV/SOF) — Exposure of interest for participants who received a LDV/SOF-based regimen in previous Gilead-sponsored chronic hepatitis C infection trials
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: Sofosbuvir/Velpatasvir (SOF/VEL) — Exposure of interest for participants who received a SOF/VEL-based regimen in previous Gilead-sponsored chronic hepatitis C infection trials
  Other Names: Epclusa®; GS-7977/GS-5816
Drug: Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX) — Exposure of interest for participants who received a SOF/VEL/VOX-based regimen in previous Gilead-sponsored chronic hepatitis C infection trials
  Other Names: Vosevi®; GS-7977/GS-5816/GS-9857

SUMMARY:
This Registry will enroll adolescent and pediatric participants who received at least one Gilead Hepatitis C Virus (HCV) direct acting antiviral (DAA) while participating in a Gilead-sponsored chronic hepatitis C clinical trial. The primary objective of this Registry is to determine the long-term safety of anti-HCV regimens in the pediatric population. Secondary objectives of this Registry are to determine whether subsequent detection of HCV RNA in participants who relapse following sustained virologic response (SVR) represents the re-emergence of pre-existing virus, the development of resistance mutations, or whether it is due to re-infection, and to characterize resistance mutations and the persistence of resistance mutations in pediatric participants who did not achieve SVR. Once enrolled, participants will be followed for up to 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Have previously participated in a Gilead-sponsored chronic hepatitis C study as an adolescent or pediatric participant and received at least one Gilead HCV direct acting antiviral
* Parent or legal guardian able to provide written informed consent OR individual is able to provide written informed consent prior to any study procedures and willing to comply with study requirements as determined by institutional review board (IRB)/independent ethics committee(IEC)/local requirements and Investigator's discretion.
* Individual is able to provide written assent, if they have the ability to read and write, as determined by IRB/IEC/local requirements and Investigator's discretion

Key Exclusion Criteria:

* Individual is currently receiving or plans to initiate a new course of hepatitis C therapy including any investigational drug or device during the course of the follow-up Registry.
* History of clinically-significant illness or any other major medical disorder that may interfere with the individual's follow-up, assessments or compliance with the protocol.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who participated in a Gilead-sponsored chronic hepatitis C study as an adolescent or pediatric participant and received at least one Gilead HCV direct acting antiviral (DAA)
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Growth data as measured by body height | Up to 5 years
Growth data as measured by body weight | Up to 5 years
Development as measured by Tanner Pubertal Stage Assessment | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (51):
- United States (27):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Div. of Research Immunology/BMT, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - UNC Pediatrics/NC Children's Hospital, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Children's Hospital, Morgantown, West Virginia
- Australia (3):
  - John Hunter Children's Hospital (JHCH), New Lambton Heights, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital, Parkville, Victoria
- Cliniques Universitaires Saint- LUC UCL, Brussels, Belgium
- Germany (2):
  - Charité Universitätsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Helios Klinikum Wuppertal, Wuppertal
- Italy (7):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria - Ospedale Pediatrico Meyer, Florence
  - Polo Universitario - L'Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero-Universitaria di Padova, Padua
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
- Auckland Clinical Studies, Auckland, New Zealand
- Poland (2):
  - Wojewódzki Szpital Obserwacyjno-Zakaźny im. Tadeusza Browicza, Klinika Chorób Zakaźnych i Hepatologii Wieku Rozwojowego, Bydgoszcz
  - MED. POLONIA Sp. z.o.o., Poznan
- Russia (4):
  - Federal Budget Institution of Science-Central Scientific and Research Institute of Epidemiology, Moscow
  - Federal Government Institution "Republican Clinical Infectious Hospital", Saint Petersburg
  - Scientific-Research Institute of Children's Infections of Federal Medico- Biological Agency, Saint Petersburg
  - Ltd Medical Company "Hepatolog", Tolyatti
- United Kingdom (4):
  - Birmingham Childrens Hospital NHS Trust, Birmingham
  - Royal Hospital for Sick Children Glasgow, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Gonzalez-Peralta RP, Wen JW, Hardikar W, Karnsakul WW, Whitworth S, Lin CH, Indolfi G, Rosenthal P, Balistreri W, Schwarz KB, Honegger JR, Zhang X, Svarovskaia EC, Suri V, Kersey K, Leung DH. Long-term efficacy and safety of sofosbuvir-based direct-acting antiviral regimens in paediatric patients with hepatitis C virus infection: an international registry study. Lancet Child Adolesc Health. 2025 Apr;9(4):248-254. doi: 10.1016/S2352-4642(25)00028-8. PMID 40113366
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-334-1113